CLINICAL TRIAL: NCT05499078
Title: Pilot Study to Assess Performance and Safety of SULFEX 13081.22 Nasal Spray in Patients With Dry or Irritated Nose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-20-F10
Record Dates: First submitted 2022-07-06; First posted 2022-08-12 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-07

CONDITIONS: Dry Nose; Nose Irritation
Keywords: Nasal Obstruction; Nasal Obstruction, Bilateral; Nasal Bleeding; Nasal Passage Irritation; Nasal Pain; Nasal Crusting; Nasal Itching; Nasal Burning; Nasal Discomfort; Sneezing; Airborne particles; Mucous Membrane
MeSH Terms: conditions — Nasal Obstruction; Epistaxis; Sneezing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SULFEX 13081.22 (Experimental): Patients with dry or irritated nose treated with SULFEX 13081.22 nasal spray for 6 days (with at least 1 spray use a day).
  Interventions: Device: SULFEX 13081.22

INTERVENTIONS:
Device: SULFEX 13081.22 — Patients with dry or irritated nose treated with SULFEX 13081.22 nasal spray for 6 days (with at least 1 spray use a day). Severity of the nasal symptoms will be compared before and 6 days after spray use on a 7-point nasal symptoms scale basis.

SUMMARY:
As the medical device is CE marked, the objective of this study is to provide performance and safety data on SULFEX 13081.22 nasal spray as close as possible to the routine care.

DETAILED DESCRIPTION:
Every day, people breathe large amounts of air which contain all kinds of particles. Nasal cavities are the first site of airway protection against airborne particles. The mucociliary apparatus (a layer of tiny moving hairs and mucus which covers the mucous membrane inside the nose) is the first line of defence of the upper airways and helps to eliminate these particles. If this defence mechanism is altered, it may cause nasosinusal damage or irritation and be unable to protect the respiratory system.

Moreover, external factors such as pollution or dry air may affect the function of the nose. The same is true for chronic and/or recurrent infections. These various factors can cause irritation or dryness of the nasal mucosa, often causing inflammation with feelings of congestion, discomfort or burning of the nasal mucosa, sometimes with bleeding or painful crusting.

SULFEX 13081.22 is a nasal spray, CE marked and commercialized since 2014. SULFEX spray soothes, restores and provides long-lasting/intense hydration of uncomfortable, painful or sore nasal mucosa caused by excessive dryness. It also contributes towards cell regeneration for faster healing and optimum relief and protects against new external attacks.The anti-reflux valve system prevents any contamination of the solution, even after the bottle has been opened, which means the formula remains 100% aseptic.

As the medical device is CE marked, the objective of this study is to provide performance and safety data on SULFEX 13081.22 nasal spray as close as possible to the routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age.
* Patient voluntarily buying the spray and using it for him/herself.
* Patient with nasal dryness and/or nasal irritation.
* Patient informed of the study, who gave its express consent (free, informed, written) before any specific procedure to the study.
* Patient meeting study's requirements regarding follow-up schedule and questionnaires filling.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient currently taking corticosteroids or antibiotics or antihistamines or Nonsteroidal anti-inflammatory drugs (NSAIDs) or topical decongestants or systemic decongestants
* Patient currently using other nasal sprays, nasal pumps, nasal irrigation/lavage device, or oils, creams or gels into the nose.
* Patient deprived of freedom or subject to legal protection measures.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Nasal symptoms severity | 6 days
  Severity of the following nasal symptoms will be compared before and 6 days after spray use on a 7-point scale basis.
  * Nasal irritation
  * Nasal dryness Performance on Irritation and Dryness will be verified if there is a decrease of at least 0.5 point on at least one of the two symptom scores between Day 0 and Day 6. This item is scaled from 0 to 3, with 0.5 increments and 3 being the worst value.

SECONDARY OUTCOMES:
Safety data on SULFEX 13081.22 nasal spray | 6 days
  To collect safety data on the SULFEX 13081.22 nasal spray after 6 days of use (with at least 1 spray use a day). Proportion of patients with at least one adverse device effect occurred between the first and the last spray use.
Performance of SULFEX 13081.22 nasal spray | 6 days
  To assess the performance of the SULFEX 13081.22 nasal spray, on the following nasal symptoms, after 6 days of use (with at least 1 spray use a day).
  * Nasal crusting
  * Nasal bleeding
  * Nasal itching
  * Nasal burning
  * Nasal obstruction
  * Nasal pain
  * Nasal discomfort
  * Sneezing
  * Reduced sense of smell
  * External nasal redness
  * External nasal swelling Performance on a particular symptom will be verified if there is a decrease of at least 0.5 point in the symptom score between Day 0 and Day 6.
  This item is scaled from 0 to 3, with 0.5 increments and 3 being the worst value.
Nasal symptoms relief/change | 6 days
  To assess nasal symptoms relief/reduction each day, from Day 0 to Day 6. Assessment of nasal symptoms mean scores at D0 / D1 / D2 / D3 / D4 / D5 and D6.
  This item is scaled from 0 to 3, with 0.5 increments and 3 being the worst value.
Onset of relief | immediate or semi-immediate
  To assess onset of relief (immediate or semi-immediate relief). Proportion of patients with immediate or semi-immediate relief.
  An immediate relief is defined as a nasal symptom improvement at 1 min or 10 min after the 1st spray use of the day. A semi-immediate relief is defined as a nasal symptom improvement at 1 hour after the 1st spray use of the day.
Duration of relief (long lasting). | 6 days
  To assess duration of relief (long lasting). This item is scaled from 0 to 3, with 0.5 increments and 3 being the worst value.
Previous nasal state of well-being assessment | 6 days
  To assess the day at which patients regained their previous nasal state of well-being (feeling of well-being). Day at which the patient regained his/her previous nasal state of well-being (feeling of well-being) + proportion of patients with an overall relief.
  This item is scaled from 0 to 3, with 0.5 increments and 3 being the worst value.
Medical device usability | 6 days
  To assess the medical device usability. assessment of the proportion of patients that would agree with each usability criteria on a 5-point scale basis.
  This item is scaled from 1 to 5, with 1 increments and 1 being the worst value.
Product attributes | 6 days
  To assess product attributes of the medical device. Assessment of proportion of patients that would agree with each product attribute on a 5-point scale basis.
  This item is scaled from 1 to 5, with 1 increments and 1 being the worst value.
Patient satisfaction | 6 days
  To assess patient satisfaction regarding the medical device. Assessment of Proportion of patients satisfied with the medical device use on a 5-point scale basis.
  * Proportion of patient liking the medical device on a 5-point scale basis + aspect that is most liked and disliked about the medical device.
  * Proportion of patients wishing to continue using the medical device on a 5-point scale basis.
  * Proportion of patients that would recommend the medical device on a 5-point scale basis.
  This item is scaled from 1 to 5, with 1 increments and 1 being the worst value.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pharmacie Lair, Vire, Normandy
  - Pharmacie Plaisance, Paris